CLINICAL TRIAL: NCT07151872
Title: A Phase II Clinical Study to Evaluate the Efficacy and Safety of QLS31905 for Injection in Combination With Chemotherapy ± QL2107 in Patients With CLDN18.2-positive Advanced Biliary Tract Cancer
Brief Title: Combination of QLS31905 and Chemotherapy ± QL2107 in Patients With CLDN18.2-positive Advanced Biliary Tract Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QLS31905-205
Record Dates: First submitted 2025-08-25; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: CLDN18.2-positive Advanced Biliary Tract Cancer
MeSH Terms: interventions — Injections; Gemcitabine; Cisplatin; Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- QLS31905 +GP (Experimental)
  Interventions: Drug: QLS31905 for Injection; Drug: Gemcitabine Hydrochloride for Injection; Drug: Cisplatin for Injection
- QLS31905 +GP+QL2107 (Experimental)
  Interventions: Drug: QLS31905 for Injection; Drug: Gemcitabine Hydrochloride for Injection; Drug: Cisplatin for Injection; Drug: QL2107 Injection
- QLS31905 +XELOX (Experimental)
  Interventions: Drug: QLS31905 for Injection; Drug: Oxaliplatin Injection; Drug: Capecitabine Tablets

INTERVENTIONS:
Drug: QLS31905 for Injection — QLS31905 for Injection
Drug: Gemcitabine Hydrochloride for Injection — Gemcitabine Hydrochloride for Injection
  Arms: QLS31905 +GP; QLS31905 +GP+QL2107
Drug: Cisplatin for Injection — Cisplatin for Injection
  Arms: QLS31905 +GP; QLS31905 +GP+QL2107
Drug: QL2107 Injection — QL2107 Injection
  Arms: QLS31905 +GP+QL2107
Drug: Oxaliplatin Injection — Oxaliplatin Injection
  Arms: QLS31905 +XELOX
Drug: Capecitabine Tablets — Capecitabine Tablets
  Arms: QLS31905 +XELOX

SUMMARY:
This is an open-label, multicenter Phase II clinical study aimed at evaluating the efficacy, safety, PK profile, and immunogenicity of QLS31905 for Injection combined with Chemotherapy ± QL2107 in Patients with CLDN18.2-positive Advanced Biliary Tract Cancer

ELIGIBILITY:
Inclusion Criteria:

* Subjects with unresectable locally advanced or metastatic Biliary Tract Cancer confirmed by histopathological or cytological examination;
* Subjects with at least one measurable lesion designated as a target lesion, as assessed by the investigator according to RECIST v1.1. Lesions that have received radiotherapy or other local treatments may be considered measurable if they demonstrate imaging PD;
* No prior systemic anti-tumor treatment for locally advanced or metastatic Biliary Tract Cancer.

Exclusion Criteria:

* Subjects with a known history of severe or repeated allergy, intolerance, or contraindication to QLS31905, QL2107, or other large molecule protein preparations, as well as Gemcitabine Hydrochloride for Injection, Cisplatin for Injection, Oxaliplatin Injection or Capecitabine Tablets and any components in their preparations;
* Subjects had other second primary malignancies within 5 years prior to the first dose;
* Subjects with clinically significant hemorrhage within 3 months before the first dose;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
ORR (Objective Response Rate) | Approximately 24 months
  ORR is defined as the proportion of participants who have a best overall response of Complete Response (CR) or Partial Response (PR) as assessed by investigator per RECIST 1.1